CLINICAL TRIAL: NCT00043030
Title: Survey Of Patient's Motivations, Perceptions, And Expectations In Phase I Clinical Trials
Brief Title: Evaluating Patient Participation in Phase I Clinical Trials
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Collaborators: National Cancer Institute (NCI) (NIH)
Other Study IDs: 020204; 02-C-0204; CDR0000069497
Record Dates: First submitted 2002-08-05; First posted 2003-01-27 (Estimated); Last update posted 2012-03-15 (Estimated); Status verified 2012-03

CONDITIONS: Psychosocial Effects of Cancer and Its Treatment; Unspecified Adult Solid Tumor, Protocol Specific
Keywords: psychosocial effects of cancer and its treatment; unspecified adult solid tumor, protocol specific
MeSH Terms: interventions — Psychiatric Rehabilitation

INTERVENTIONS:
Procedure: psychosocial assessment and care

SUMMARY:
RATIONALE: Understanding why patients participate in a phase I clinical trial may help doctors plan better treatment for cancer.

PURPOSE: This clinical trial is studying to determine the reasons for participation, perceptions, and expectations of patients receiving treatment for cancer in phase I clinical trials.

DETAILED DESCRIPTION:
OBJECTIVES:

* Describe the motivations, perceptions, and expectations of patients enrolled in a phase I clinical trial.
* Assess the influence of age, education, and gender upon the perception of these patients.
* Compare the difference in perceptions, motivations, and expectations of patients who have previously participated in a phase I clinical trial vs those who have not.
* Determine whether patients' perceptions, motivations, and expectations change while enrolled in a phase I clinical trial.
* Validate an interviewer-administered tool measuring the perceptions, motivations, and expectations of these patients.
* Assess patients' perception of the information they were given while enrolled in a phase I clinical trial.

OUTLINE: Patients are interviewed over the phone to evaluate their perceptions, motivations, and expectations of phase I clinical trials. Patients complete a questionnaire comprising 24 questions over 30-45 minutes. Interviews are conducted within 1 week after enrolling in a phase I clinical trial (prior to the first dose of study agent) and then again 2 months later (or at the time the patient stops treatment). The first 10 patients enrolled complete an additional 6 questions over 15 minutes during the first interview to validate the questionnaire, but do not complete a second interview.

PROJECTED ACCRUAL: A total of 120 patients will be accrued for this study within 1 year.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Enrolled in a phase I clinical trial within the past week

  * Signed an informed consent for a phase I trial

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* Not specified

Life expectancy

* Not specified

Hematopoietic

* Not specified

Hepatic

* Not specified

Renal

* Not specified

Other

* Able to follow basic verbal instructions as witnessed by the investigator or a representative
* Able to understand and speak English as determined by the investigator or a representative
* Access to a telephone

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* Not specified

Endocrine therapy

* Not specified

Radiotherapy

* Not specified

Surgery

* Not specified

Other

* Prior participation in a phase I clinical trial allowed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2002-06; Primary Completion 2006-12 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
Patients' perceptions, motivations, and expectations as assessed by survey prior to and 2 months after enrollment on a phase I clinical trial

SECONDARY OUTCOMES:
Influence of age and education on perception as assessed by survey prior to and 2 months after enrollment on a phase I clinical trial
Compare difference between patients who have and who have not previously participated in phase I clinical trials as assessed by survey prior to and 2 months after enrollment on a phase I clinical trial
Changes in patients' perceptions, motivations, and expectations as assessed by survey prior to and 2 months after enrollment on a phase I clinical trial
Validate measurement of patients' perceptions, motivations, and expectations as assessed by survey prior to and 2 months after enrollment on a phase I clinical trial
Patient's perceptions of information given as assessed by survey prior to and 2 months after enrollment on a phase I clinical trial
Influence of gender upon perception as assessed by survey prior to and 2 months after enrollment on a phase I clinical trial

CONTACTS AND LOCATIONS:
Overall Officials: Arlene Berman, RN, MS, OCN, Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- Warren Grant Magnuson Clinical Center - NCI Clinical Studies Support, Bethesda, Maryland, United States